CLINICAL TRIAL: NCT04735744
Title: Evaluation of Allied Healthcare in Patients Recovering From COVID-19
Acronym: ParaCOV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: ParaCOV
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Allied Health Professionals; Primary Care; Retrospective Cohort; PROMs; Performance Measures; Prospective Cohort; National Dutch Program
Keywords: Covid19; Allied health professionals; primary care; PROMs
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: Allied health professionals (i.e., dietitians, exercise therapists, physical therapists, occupational therapists and speech and language therapists) that treat patients recovering from COVID-19 in Dutch primary care
  Interventions: Other: Patients recovering from COVID19 receive usual care by allied health professionals
- Retrospective cohort: Allied health professionals (i.e., dietitians, exercise therapists, physical therapists, occupational therapists and speech and language therapists) that have been treated patients recovering from COVID-19 in Dutch primary care
  Interventions: Other: Patients recovering from COVID19 receive usual care by allied health professionals

INTERVENTIONS:
Other: Patients recovering from COVID19 receive usual care by allied health professionals — We will not develop specific interventions for this prospective observational cohort study. The care provided by allied health professionals in daily practice are based on recommendations published by the professional bodies of allied health professionals and on the interdisciplinary guidance developed by the LAN. All allied health professionals are working according to these recommendations. Dissemination of these recommendations is done by the professional bodies of the allied health professionals. Given the observational nature of our study, no additional implementation strategies will be employed to stimulate this care by the research group.

SUMMARY:
SUMMARY Rationale: Allied health professionals (i.e., dietitians, exercise therapists, physical therapists, occupational therapists and speech and language therapists) might play an important role in the recovery of patients with COVID-19 who experience limitations in daily physical functioning and participation. However, the evidence base for allied healthcare in patients with COVID-19 has yet to be established. To facilitate care for people recovering from COVID-19 and to establish this evidence base, the Dutch ministry has created a temporary regulation for primary care allied healthcare specifically for patients with COVID-19.

Objective: This study is setup alongside the temporary regulation and aims to evaluate the longitudinal recovery trajectories and related costs of patients who visited a primary care allied healthcare professional for the management of severe symptoms and activity limitations and/or participation restrictions related to COVID-19.

Study design: Prospective cohort study. Study population: 1,315 adult patients recovering from COVID-19 with severe symptoms and activity limitations and/or participation restrictions, and who are referred to a primary care allied health professional by a general practitioner or medical specialist within four months of the start of the disease will be eligible for this study.

Intervention (if applicable): Although the nature of this study is non-experimental, the allied healthcare intervention can be considered experimental due to the novelty of the disease.

Main study parameters/endpoints: The primary outcome domain of this study is participation measured with the Utrechtse Schaal voor Revalidatie - Participatie (USER-P). The primary endpoint is set at 6 months. A 5 point difference will be considered clinically relevant for patients with COVID-19.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no specific risks involved with participation in this study, as it entails the completion of questionnaires over the timeframe of one year (at the start of the treatment, the end of the treatment, 3 months, 6 months, 9 months and 12 months). The load of the survey will be highest at months 3, 6 and 12 with a total of 74 survey items. Input from patient representatives suggested that this number of items was feasible, especially because participants are allowed to complete the survey over a number of days. Finally, none of the items in the survey are considered emotionally distressing. The prescribed interventions are conform the recommendations of the best available evidence and are in line with usual allied healthcare interventions. Therefore, risks are likely to be negligible conform usual allied healthcare.

ELIGIBILITY:
Inclusion Criteria:

Adult patients

* recovering from COVID-19 with severe symptoms and activity limitations and/or participation restrictions, and;
* who are referred to a primary care allied health professional by a general practitioner or medical specialist within four months of the start of the disease; will be eligible for this study. The need for referring the patient to an allied health professional will be judged by the primary care physician or medical specialist. Criteria for referral are described in guidance published by the Long Alliantie Nederland (LAN) with recommendations for treatment of post-COVID-19-patients: the COVID-19 Associated Syndrome (CAS) (Chapters 3.3 and 4).

http://www.longalliantie.nl/files/2515/9359/4621/Handreiking_voor_de_zorg.pdf

Exclusion Criteria:

Adult patients:

- receiving palliative care; are excluded from this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients of 18 year and older recovering from COVID-19 with severe symptoms and activity limitations and/or participation restrictions, who are referred to a primary care allied health professional* by a general practitioner or medical specialist are deemed eligible for this study.
  *Allied health professionals relevant to this study are: Dietitians, Exercise Therapists, Occupational Therapists, Physical Therapists, and Speech and Language Therapists working in primary care in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 1441 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-07-17 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Participation | Baseline (T0)
  Measured with the Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P) (32 items)
Participation | 3 months (T1)
  Measured with the Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P) (32 items)
Participation | 6 months (T2)
  Measured with the Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P) (32 items)
Participation | 12 months (T3)
  Measured with the Utrecht Scale for Evaluation of Rehabilitation Participation (USER-P) (32 items)
Quality of life measured with EQ-5D-5L | Baseline (T0)
  Measured with the EuroQol five-dimensional questionnaire (EQ-5D-5L) (5 items)
Quality of life measured with EQ-5D-5L | 3 months (T1)
  Measured with the EuroQol five-dimensional questionnaire (EQ-5D-5L) (5 items)
Quality of life measured with EQ-5D-5L | 6 months (T2)
  Measured with the EuroQol five-dimensional questionnaire (EQ-5D-5L) (5 items)
Quality of life measured with EQ-5D-5L | 12 months (T3)
  Measured with the EuroQol five-dimensional questionnaire (EQ-5D-5L) (5 items)
Fatigue | Baseline (T0)
  Measured with the Fatigue Severity Scale (FSS)
Fatigue | 3 months (T1)
  Measured with the Fatigue Severity Scale (FSS)
Fatigue | 6 months (T2)
  Measured with the Fatigue Severity Scale (FSS)
Fatigue | 12 months (T3)
  Measured with the Fatigue Severity Scale (FSS)
Physical functioning | Baseline (T0)
  PROMIS Physical Functioning Short Form 10b (10 items).
Physical functioning | 3 months (T1)
  PROMIS Physical Functioning Short Form 10b (10 items).
Physical functioning | 6 months (T2)
  PROMIS Physical Functioning Short Form 10b (10 items).
Physical functioning | 12 months (T3)
  PROMIS Physical Functioning Short Form 10b (10 items).
Costs | Baseline (T0)
  will be measured using a cost questionnaire (18 items)
Costs | 3 months (T1)
  will be measured using a cost questionnaire (18 items)
Costs | 6 months (T2)
  will be measured using a cost questionnaire (18 items)
Costs | 9 months (T3)
  will be measured using a cost questionnaire (18 items)
Costs | 12 months (T4)
  will be measured using a cost questionnaire (18 items)
Patient Specific Activities | baseline (T0) as part of usual care
  measured with the Patient Specific Complaints (PSC)
Patient Specific Activities | end of the treatment as part of usual care (average of 6 months)
  measured with the Patient Specific Complaints (PSC)
Nutritional Status | baseline (T0) as part of usual care
  measured with the BMI (weight and height)
Nutritional Status | end of the treatment as part of usual care (average of 6 months)
  measured with the BMI (weight and height)
Global Assessment | baseline (T0) as part of usual care
  measured with the PG-SGA short form weight history, food intake, symptoms, activities and function).
Global Assessment | end of the treatment as part of usual care (average of 6 months)
  measured with the PG-SGA short form weight history, food intake, symptoms, activities and function).
Voice Problems | baseline (T0) as part of usual care
  measured with Voice Handicap Index (VHI)
Voice Problems | end of the treatment as part of usual care (average of 6 months)
  measured with Voice Handicap Index (VHI)
Swallowing Problems | baseline (T0) as part of usual care
  Dysphagia Handicap Index (DHI).
Swallowing Problems | end of the treatment as part of usual care (average of 6 months)
  Dysphagia Handicap Index (DHI).
Patient Specific Activities | baseline (T0) as part of usual care
  measured with the Canadian Occupational Performance Measure (COPM)
Patient Specific Activities | end of the treatment as part of usual care (average of 6 months)
  measured with the Canadian Occupational Performance Measure (COPM)
Activities | baseline (T0) as part of usual care
  measured with the PRO-ergo
Activities | end of the treatment as part of usual care (average of 6 months)
  measured with the PRO-ergo

SECONDARY OUTCOMES:
Exercise capacity | baseline (T0) as part of usual care
  6 Minute Walk Test (6MWT)
Exercise capacity | end of the treatment as part of usual care (average of 6 months)
  6 Minute Walk Test (6MWT)
Exercise capacity | baseline (T0) as part of usual care
  Short Physical Performance Battery (SPPB)
Exercise capacity | end of the treatment as part of usual care (average of 6 months)
  Short Physical Performance Battery (SPPB)
Quadriceps strength | baseline (T0) as part of usual care
  with a hand dynamometer.
Quadriceps strength | end of the treatment as part of usual care (average of 6 months)
  with a hand dynamometer.
Hand grip strength | baseline (T0) as part of usual care
  with a hand dynamometer.
Hand grip strength | end of the treatment as part of usual care (average of 6 months)
  with a hand dynamometer.
Bioimpedance (BIA | baseline (T0) as part of usual care
Bioimpedance (BIA | end of the treatment as part of usual care (average of 6 months)
VAS-appetite, taste and smell | baseline (T0) as part of usual care
VAS-appetite, taste and smell | end of the treatment as part of usual care (average of 6 months)
Dietary goal attainment | baseline (T0) as part of usual care
Dietary goal attainment | end of the treatment as part of usual care (average of 6 months)
Liquid medical nutrition | baseline (T0) as part of usual care
Liquid medical nutrition | end of the treatment as part of usual care (average of 6 months)
Sarcopenia | baseline (T0) as part of usual care
  measured with the SARC-F
Sarcopenia | end of the treatment as part of usual care (average of 6 months)
  measured with the SARC-F
Types of Stool | baseline (T0) as part of usual care
  measured with the Bristol Stool Chart (BCS)
Types of Stool | end of the treatment as part of usual care (average of 6 months)
  measured with the Bristol Stool Chart (BCS)
Voice Problems | baseline (T0) as part of usual care
  measured with Maximum Phonation Time (MPT)
Voice Problems | end of the treatment as part of usual care (average of 6 months)
  measured with Maximum Phonation Time (MPT)
Swallowing Problems | baseline (T0) as part of usual care
  measured with Maximum Swallowing Speed (MSP)
Swallowing Problems | end of the treatment as part of usual care (average of 6 months)
  measured with Maximum Swallowing Speed (MSP)
Physical Functioning | baseline (T0) as part of usual care
  measured with the Assessment of Motor and Process Skills (AMPS)
Physical Functioning | end of the treatment as part of usual care (average of 6 months)
  measured with the Assessment of Motor and Process Skills (AMPS)
Cognitive Functioning | baseline (T0) as part of usual care
  measured with the Cognitive Complaints - Participation (CoCo-P)
Cognitive Functioning | end of the treatment as part of usual care (average of 6 months)
  measured with the Cognitive Complaints - Participation (CoCo-P)

CONTACTS AND LOCATIONS:
Overall Officials: Philip van der Wees, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Slotegraaf AI, Kruizenga HM, Gerards MHG, Verburg AC, Hoogeboom TJ, de van der Schueren MAE; Dutch Consortium Allied Healthcare COVID-19. Risk of poor nutritional status and nutrition-related complaints in individuals attending a primary care dietitian after a COVID-19 infection: A prospective cohort study. Nutr Diet. 2025 Apr;82(2):172-185. doi: 10.1111/1747-0080.12905. Epub 2024 Oct 21. PMID 39429046
- [Derived] Ben AJ, Verburg AC, Maas ET, Hoogeboom TJ, Gerards MHG, Slotegraaf AI, Cup EHC, Schaafsma F, W J G Ostelo R, van Dongen JM; Dutch Consortium Allied Healthcare COVID-19, ParaCOV cohort study. Work Trajectories of Patients With Persistent Complaints After a COVID-19 Infection Receiving Allied Healthcare in the Netherlands: A Secondary Analysis of the ParaCOV Cohort. J Occup Environ Med. 2024 Dec 1;66(12):993-999. doi: 10.1097/JOM.0000000000003240. Epub 2024 Oct 10. PMID 39393926
- [Derived] Gerards MHG, Slotegraaf AI, Verburg AC, Kruizenga HM, Cup EHC, Kalf JG, Lenssen AF, Meijer WM, Ben AJ, van Dongen JM, de van der Schueren MAE, Graff MJL, Akkermans RP, van der Wees PJ, Hoogeboom TJ; Dutch Consortium Allied Healthcare COVID-19. One-year evaluation of people recovering from COVID-19 receiving allied primary healthcare: A nationwide prospective cohort study. Ann Phys Rehabil Med. 2024 Oct;67(7):101874. doi: 10.1016/j.rehab.2024.101874. Epub 2024 Aug 21. PMID 39173549
- [Derived] Slotegraaf AI, de Kruif AJTCM, Agasi-Idenburg CS, van Oers SMD, Ronteltap A, Veenhof C, Gerards MHG, Verburg AC, Hoogeboom TJ, de van der Schueren MAE; Dutch Consortium Allied Healthcare COVID-19. Understanding recovery of people recovering from COVID-19 receiving treatment from primary care allied health professionals: a mixed-methods study. Disabil Rehabil. 2024 Dec;46(24):5798-5807. doi: 10.1080/09638288.2024.2311330. Epub 2024 Feb 6. PMID 38318773
- [Derived] Slotegraaf AI, Gerards MHG, Verburg AC, de van der Schueren MAE, Kruizenga HM, Graff MJL, Cup EHC, Kalf JG, Lenssen AF, Meijer WM, Kool RA, de Bie RA, van der Wees PJ, Hoogeboom TJ; Dutch Consortium Allied Healthcare COVID-19. Evaluation of Primary Allied Health Care in Patients Recovering From COVID-19 at 6-Month Follow-up: Dutch Nationwide Prospective Cohort Study. JMIR Public Health Surveill. 2023 Oct 20;9:e44155. doi: 10.2196/44155. PMID 37862083